CLINICAL TRIAL: NCT05707533
Title: Vaginal Adventitia Reserved and Anatomical Implant Technique of Transvaginal Mesh Procedure for Pelvic Organ Prolapse: 13-year Surgical Results With 589 Cases
Brief Title: Vaginal Adventitia Reserved and Anatomical Implant Technique of Transvaginal Mesh Procedure for Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, De-yi Luo, Prof., West China Hospital
Other Study IDs: 2021833
Record Dates: First submitted 2022-12-18; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Complication; Transvaginal Mesh Procedure
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Cefoxitin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients underwent TVM using the Vaginal Adventitia Reserved and Anatomical Implant Technique: Patients with pelvic organ prolapse who underwent TVM using the Vaginal Adventitia Reserved and Anatomical Implant Technique between June 2008 and December 2020
  Interventions: Procedure: TVM using the Vaginal Adventitia Reserved and Anatomical Implant Technique

INTERVENTIONS:
Procedure: TVM using the Vaginal Adventitia Reserved and Anatomical Implant Technique — The Transvaginal mesh procedure with Vaginal Adventitia Reserved and Anatomical Implant Technique for the treatment of POP. The Cefoxitin Injection Solution was used for Prophylactic antibiotics
  Other Names: Cefoxitin

SUMMARY:
After obtaining an institutional ethics approval (#2021833), the investigators retrospectively reviewed patients with Pelvic organ prolapse (POP) who underwent Transvaginal Mesh (TVM) in their hospital during June 2008 and December 2020. The goal of this observational study is to introduce the Vaginal Adventitia Reserved and Anatomical Implant Technique in Transvaginal mesh surgery, and to report long term efficacy and safety results of this technique. The main questions it aims to answer are:

* How to reduce the potential risk of mesh-related complications when performing TVM?
* How effective is the use of the Vaginal Adventitia Reserved and Anatomical Implant Technique when performing TVM? Participants will be asked to fill the Pelvic Floor Distress Inventory (PFDI-20) at final follow-up, and the Prosthesis/Graft Complication Classification Code was used to record the mesh-related complications.

DETAILED DESCRIPTION:
Patients and materials The investigators retrospective reviewed consecutive patients with stage II to IV Pelvic organ prolapse (POP) who underwent Transvaginal Mesh (TVM) at their center from June 2008 to December 2020. The Vaginal Adventitia Reserved and Anatomical Implant Technique was performed on all patients. Informed consent was obtained from all included patients. Approval was obtained from the institutional ethics committee of our hospital (West China Hospital, Sichuan University).

The pre-cut mesh kits including Gynecare Prolift® (Ethicon, Sommerville, NJ, USA), Perigee (AMS, Minnetonka, MN, USA), and Gynecare Prosima® (Ethicon, Sommerville, NJ, USA) and self-cut mesh Gynemesh (Ethicon, Sommerville, NJ, USA) were applied for transvaginal mesh repair in this study. Surgery was performed by an experienced surgeon (Dr. HS), utilizing the vaginal adventitia reserved and anatomical implant technique.

Outcome measures The effect of operation was assessed using both objective and subjective measures. The objective assessment (anatomic assessment) of success was that the nadir of prolapse never reached the point 0 (the level of hymen). The subjective assessment of success was the absence of prolapse symptoms. Chinese version of the Pelvic Floor Distress Inventory (PFDI-20) was also utilized for assessing the outcomes. Prosthesis/Graft Complication Classification Code was used to record the mesh-related complications.

Data analysis Statistical analysis was performed via the commercially available statistical package (SPSS) 22.0 for Windows (SPSS, Chicago, IL, USA). Categorical variables were represented using frequency and percentages and compared using the chi-square test. Continuous variables in accord with normal distribution were described using means and standard deviations (SDs) and analyzed using the Student's t-test. Statistical significance was defined at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yr
* Clinical diagnosis of pelvic organ prolapse
* Pelvic organ prolapse-quantification (POP-Q) > II stage
* Patients underwent TVM using the Vaginal Adventitia Reserved and Anatomical Implant Technique

Exclusion Criteria:

* Patients who refused to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with POP who underwent TVM using the Vaginal Adventitia Reserved and Anatomical Implant Technique at the investigators' center from June 2008 to December 2020.
Sampling Method: Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse-Quantification (POP-Q) scores | The time frame was from the date of surgery to the date of final follow-up, ranging from 9 to 156 months.
  The POP-Q system was used to assess the pelvic organ prolapse
complication | The time frame was from the date of surgery to the date of final follow-up, ranging from 9 to 156 months.
  Prosthesis/Graft Complication Classification Code was used to record the mesh-related complications
Pelvic Floor Distress Inventory (PFDI-20) scores | The time frame was from the date of surgery to the date of final follow-up, ranging from 9 to 156 months.
  The PFDI-20 was used to assess pelvic floor symptoms and associated bother and has 3 subscales: the pelvic organ prolapse distress inventory (POPDI)(0-300); the colorectal-anal distress inventory (CRADI)(0-400); and the urinary distress inventory (UDI)(0-300). Higher scores indicted greater symptom bother.
Female Sexual Function Index (FSFI) scores | The time frame was from the date of surgery to the date of final follow-up, ranging from 9 to 156 months.
  FSFI was used to assess the sexual function, which was a validated questionnaire comprised of 19 items. FSFI's total score ranged from 2 to 36; the higher the score, the severer the sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-min Li, PhD., Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided